CLINICAL TRIAL: NCT07267754
Title: Uterine Interstitial Myolisis and Oocytes Retrieval in Single Step: a Pilot Study
Acronym: UIMandOPU
Status: Not yet recruiting | Type: Observational
Sponsor: San Carlo Public Hospital, Potenza, Italy (Other)
Responsible Party: Principal Investigator, Assunta Iuliano, MD, Medical Doctor, San Carlo Public Hospital, Potenza, Italy
Other Study IDs: San Carlo PH; Comitato Etico Unico Regionale (Other: San Carlo Public Hospital, Potenza-Italy)
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy Rate IVF; Clinical Pregnancy Rate; Live Birth Rate
Keywords: Oocyte retrieval; Interstitial myolysis; Assisted Reproductive Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- infertile patients undergoing oocyte retrieval affected by uterine myomatosis: Women affected by any form of infertility aged between 18 and 45 years with uterine myomatosis who are undergoing oocyte retrieval

SUMMARY:
The aim of this observational cohort study is to evaluate the pregnancy rate, the ongoing pregnancy rate and the live birth rate of infertile women aged between 18 and 45 years who undergo a single surgical step of oocyte retrieval and uterine interstitial myolisis .

The main questions of these study are:

1. What is the chances of a positive pregnancy test and what is the chances of live birth for women who undergo oocyte retrieval and interstitial myolysis in a single surgical step?
2. Are there any complications associated with performing the two surgical techniques at the same time? Researchers will calculate IVF/ICSI outcomes after embryotransfer of vitrified blastocystis obtained after oocyte retrieval and subsequent interstitial myolysis.

Women undergoing oocyte retrieval will agree to undergo oocyte retrieval and interstitial myolysis at the same time, to freeze their blastocysts and to transfer them into the uterus after 6 months

ELIGIBILITY:
Inclusion Criteria:

Infertile women with uterine fibroids who need to undergo oocytes retrieval between 18 and 45years old

Exclusion Criteria:

Fertile woman with uterine fibroids Fertile women without uterine fibroids Women under 18 years old Woman over 45 years old

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile women with uterine fibroids who need to undergo oocytes retrieval between 18 and 45years old
Study Population: Infertile women between 18 and 45 yearsvold whith uterine fibroids who need to undergo oocyte retrieval at the "San Carlo" Medically Assisted Reproduction Center - Potenza, Italy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Chance of pregnancy after frozen embryotransfer | From the transfer of the thawed blastocyst to the birth of the baby. 18 months
  The researchers' primary objective is to calculate the pregnancy rate, miscarrage rate and live birth rate of the number of embryo transfers performed in the patients enrolled in the study.
  The pregnancy rate % per embryo transfer is a mesure of success of an embryo transfer procedure and it is calculated as follow: (number of clinical pregnancy/number of embryo trasnfer) x 100.
  The miscarriage %per embryo transfer is a measure of the risk of miscarrage following transfer procedure and it is calulated as follows: ( number of miscarrage/number of clinical pregnancies) x 100.
  The live birth rate % per embryo transfer is a measure of the success of an embryo transfer procedure in achieving a live birth and it is calculated as follows: ( number of live biths/number of embryo transfer) x 100.
IVF/ICSI outcome | 18 month
  Il tasso di gravidanza per trasferimento di embrioni è calcolato come segue: (numero di gravidanze cliniche/numero di trasferimento di embrioni) x 100. L'aborto spontaneo per trasferimento di embrioni è una misura del rischio di aborto spontaneo ed è calcolato come segue: (numero di aborti spontanei/numero di gravidanze cliniche) x 100.
  Il tasso di nati vivi per trasferimento di embrioni è una misura del successo di una procedura di trasferimento di embrioni nel raggiungimento di un parto vivo ed è calcolato come segue: (numero di nati vivi/numero di trasferimenti di embrioni) x 100.
Pregnancy Rate | 18 months after oocytes retrieval and interstitial myolysis
  (Number of clinical pregnancies/ Number of embryo transfers) x 100
Post surgical pelvic organ injury | 30 days
  Post surgical pelvic organ injury refers to any structural or functional damage to the organs within the pelvic cavity ( such as the bladder, uterus, ovaries, rectum or neurovascular structures) that occurs as a direct result of a surgical procedure. This injury may manifest as perforation, laceration, devascularization or impaired organ function and is diagnosed based on clinicalsigns, imaging or intraoperative findings
miscarriage rate | 18 months
  Number of miscarriages ( spntaneous abortions)/Number of clinicla pregnancies( x 100
Live Birth Rate | 18 months
  /Number of live births/ Number of embryo transfers ) x 100

SECONDARY OUTCOMES:
Post- surgical bleeding | 30 days
  Post surgical bleeding is a substantial loss ofl blood after oocytes retrieval or after interstial myolisis, involving the loss of at lest one gram of hemoglobin
Post surgical sepsis | 30 days
  Post surgical sepsis is a life-threatening systemic infection that develops within 30 days after a surgical procedure. It is characterzed by a dysregulatedhost response to infection, leading to organ dysfuncyion or failure. The condition requires prompt recognition, source control and broad-spectrum antimicrobial therapy to improve outcome

CONTACTS AND LOCATIONS:
Overall Officials: Assunta Iuliano, Principal Investigator, Principal Investigator — San Carlo Public Hospital, Potenza, Italy
Locations (1):
- San Carlo Public Hospital, Potenza -Italy, Potenza, PZ, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bing-song Z, Jing Z, Zhi-Yu H, Chang-tao X, Rui-fang X, Xiu-mei L, Hui L. Unplanned pregnancy after ultrasound-guided percutaneous microwave ablation of uterine fibroids: A follow-up study. Sci Rep. 2016 Jan 6;6:18924. doi: 10.1038/srep18924. PMID 26733265
- [Background] Beermann M, Jonsdottir G, Cronisoe A, Hasselrot K, Kopp Kallner H. Long term follow-up of uterine fibroids treated with microwave ablation: an up to 3-year observational study of volume, regrowth, and symptoms. Int J Hyperthermia. 2022;39(1):1158-1163. doi: 10.1080/02656736.2022.2109764. PMID 36049885
- [Background] Jonsdottir G, Beermann M, Lanz E, Nikodell A, Cronsioe A, Hasselrot K, Kopp-Kallner H. Ultrasound guided microwave ablation treatment of uterine fibroids: Clinical response and patient acceptability. Acta Obstet Gynecol Scand. 2025 Feb;104(2):350-356. doi: 10.1111/aogs.15041. Epub 2024 Dec 19. PMID 39697096
- [Background] Ahmad F, Khan AI, Asif A, Ahmed S, Nisar M, Fatima E, Khan F, Razzaq A, Tahir A, Khalid AR, Azeemuddin M. Clinical Efficacy of Percutaneous Microwave Ablation in Treating Uterine Fibroids: A Comprehensive Systematic Review and Meta-Analysis. Eur J Obstet Gynecol Reprod Biol. 2025 Jun;310:113954. doi: 10.1016/j.ejogrb.2025.113954. Epub 2025 Apr 5. PMID 40209488
- See also: Related Info — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=&cad=rja&uact=8&ved=2ahUKEwjisL_U0a6QAxV2nf0HHSfTJfwQFnoECEYQAQ&url=https%3A%2F%2Fwww.ospedalesancarlo.it%2F&usg=AOvVaw0TLuGeEjLiU7bYLeabS_GP&opi=89978449